CLINICAL TRIAL: NCT04581915
Title: A Pragmatic, Individually Randomised, Double-blind, Placebo-controlled Trial of Triazavirin (TZV) for the Treatment of Mild-moderate SARS-CoV-2 Infection A Phase II and III Clinical Trial
Brief Title: PHRU CoV01 A Trial of Triazavirin (TZV) for the Treatment of Mild-moderate COVID-19
Acronym: PHRUCov01
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: DSMB report
Sponsor: Wits Health Consortium (Pty) Ltd (Other)
Collaborators: PharmaCentrix (Pty) Ltd (Unknown); Perinatal HIV Research Unit of the University of the Witswatersrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PHRU CoV01
Record Dates: First submitted 2020-09-16; First posted 2020-10-09 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2020-10

CONDITIONS: Covid19
Keywords: SARS CoV2; Triazavirin; Novel anti-viral agent
MeSH Terms: conditions — COVID-19 | interventions — riamilovir

STUDY DESIGN:
Intervention Model Description: Participants are assigned to an interventional group or a placebo group after randomisation in parallel for the duration of the study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Pharmacists
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional (Experimental): Participants to receive Triazavirin 250mg po 8 hourly for 5 days
  Interventions: Drug: Triazavirin (Riamilovir)
- Control (Placebo Comparator): Participants to receive placebo po 8 hourly for 5 days
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Triazavirin (Riamilovir) — Capsule - 250mg 8 hourly po
  Arms: Interventional
Other: Placebo — Placebo capsule
  Arms: Control

SUMMARY:
A) Phase II: Early viral responses to triazavirin In hospitalised patients with mild-moderate COVID-19, in addition to standard of care therapy, treatment with triazavirin 250mg three times daily for five days, the slope of increase of the Ct values of serial nasopharyngeal swabs to 12 days after initiation of treatment will be ≥24% higher than in hospitalised patients receiving standard of care treatment only.

B) Phase III: Efficacy of triazavirin to improve clinical outcomes In hospitalised patients with mild-moderate laboratory proven COVID-19, in addition to standard of care therapy, treatment with triazavirin 250mg three times daily for five days will reduce a composite outcome - death; ICU admission or mechanical ventilation; or prolonged duration of admission- by ≥29% when compared to the composite outcome in hospitalised patients receiving standard of care therapy only.

DETAILED DESCRIPTION:
Design: This will be a two-site, iterative, double-blinded, randomized, placebo controlled, 2-arm, phase II and III superiority trial. Participants will be randomised 1:1 to each arm. The first part of the trial will recruit 64 evaluable patients to validate a biological effect of triazavirin on SARS-CoV-2. If triazavirin indeed has a demonstrable effect, the trial will continue to randomise another 316 evaluable participants to ascertain if there is a clinical benefit.

Participants: Three hundred and eighty evaluable patients with newly diagnosed, laboratory confirmed, mild-moderate (including asymptomatic) SARS-CoV-2 infection. Men and women will be recruited in a ratio of 3:2.

Study sites: Tshepong Provincial Hospitals in NW Province. Field Hospitals in Gauteng (NASREC) and North West (West Vaal) will be included if possible.

Study Duration: Follow up will be approximately 32 days; the total duration of from recruitment of first patients to last follow follow up visit is 15 months.

Population: Adult in-patients, ≥18 years and older, with a recent diagnostic test positive for SARS-CoV-2. Men and women will be recruited, in a ratio of 3:2.

Intervention: After verbal informed consent is provided, participants will be randomly assigned to receive either five days of triazavirin 250mg p.o three times daily, or placebo at the same dosing schedule, in addition to standard of care therapy prescribed by the attending physicians.

Primary Objectives:

To ascertain whether a 5-day course of TZV (250mg taken orally three times per day) in addition to standard of care treatment for in-patients with mild-moderate disease caused by SARS-Cov-2 is effective in:

A. Enhancing the rate of viral clearance from the nasopharynx compared to placebo.

B. To demonstrate a favourable outcome in the intervention arm compared to placebo arm using a composite clinical outcome that consists of the earliest occurrence of any of the following:

1. Death
2. Admission to ICU or mechanical ventilation required (continuous positive airway pressure, high flow nasal oxygen or intubation);
3. Prolonged duration of admission lasting >14 days (this includes patients who are discharged and re-admitted within 48 hours of leaving the hospital).

C. To ascertain safety and tolerability of the investigational drug TZV

Secondary objectives:

1. To compare time to the first of two consecutive nasopharyngeal swabs that are negative for SARS-CoV-2 between the arms.
2. To compare the proportion of participants whose nasopharyngeal swabs are negative for SARS-CoV-2 two days after the end of study treatment.
3. To compare symptom reduction and improvement in clinical measures between arms
4. To compare efficacy of nasopharyngeal swabs with salivary specimens in assessing viral responses to treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥18 years of age, who have a clinical presentation suggestive of COVID-19, or who have had a molecular laboratory assay that confirms SARS-CoV-2 infection that was collected prior to the first dose of study treatment.
2. Patients with mild to moderate COVID-19 who need admission and may require oxygen at admission but not yet requiring escalation of oxygen therapy to CPAP, high flow nasal oxygen or intubation. We will not include patients with laboratory confirmation of SARS-CoV-2 who report no symptoms at all.
3. Able to provide own consent
4. Willing to have HIV test - unless already has clinical documentation of HIV infection (as evidenced by a HIV rapid test result during the admission, or any one of the following: a positive HIV ELISA assay; an ART prescription; a pill container for ART with the patient's name; a hard copy or an electronic viral load result that includes the patient's name showing detectable HIV copies; clinical documentation of HIV sero-positivity included in the medical record)
5. Randomisation must occur within 48 hours of first COVID-19 diagnosis during the current illness.

Exclusion Criteria:

1. Women who are pregnant or breastfeeding at the time of enrolment
2. Weight <40kg.
3. Evidence of current liver disease (AST/ALT >3x ULN ; total bilirubin>3xULN or prior history of cirrhosis or other chronic liver disease)
4. Renal dysfunction as evidenced by an estimated glomerular filtration rate (eGFR) <60ml/min, or prior/current diagnosis of chronic kidney disease.
5. Prior receipt of any treatment with putative or proven anti-SARS-Cov-2 activity apart from the following: chloroquine, hydroxychloroquine, or ritonavir/lopinavir initiated no more than 12 hours prior to first receipt of TZV/placebo for this trial. Antiretrovirals initiated prior to admission as treatment for HIV, supportive, steroidal and non-steroidal anti-inflammatory, or anti-pyretic treatments are allowed.
6. Indication for immediate initiation of antiretroviral therapy in HIV-infected patients, who are unable to delay ART initiation or re-initiation until the treatment phase of this study is complete.
7. Permanently lives or works more than 120km from the hospital where recruited
8. Unable to provide own consent
9. In the opinion of either the attending doctor, or a study investigator that the patient is not a candidate for a clinical trial
10. Receipt of anti-epileptic medication, warfarin or TB treatment at the time of recruitment or during the receipt of trial treatment.
11. Enrolled currently in a trial of novel preventive treatment or treatment of SARS-CoV-2.
12. Potential participants who are investigational site staff members, or relatives of a site staff member, or those who are employees of PharmaCentrix involved in the conduct of the trial.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2020-09-08 (Actual); Primary Completion 2021-04-20 (Actual); Study Completion 2021-04-20 (Actual)

PRIMARY OUTCOMES:
To compare the slope of cycle threshold(Ct) values of nasopharyngeal swabs in people receiving Triazavirin versus placebo | 11 days per patient
  To ascertain that indeed there is a biological effect of Triazavirin, we will compare slope of cycle threshold (Ct) values of nasopharyngeal swabs taken from all patients in the Phase II part of the trial. We require at least a 24% difference in slope.
To assess the proportion of patients who progress to severe COVID-19 and the proportion who need ICU or die. | 1 month per patient
  We have selected a composite measure including three adverse outcomes, all of which have serious implications for the patient and the health system. We will combine: deaths; ICU admissions or mechanical ventilation; and prolonged hospital stays -defined in this study as >14 days.
To determine the proportion of patients who develop grade 3 or grade 4 adverse events on treatment | 1 month per patient
  We will compare rates of grade 3 and worse adverse events that occur whilst on treatment, and for up to 30 days after randomisation. We will also report on tolerability, by comparing the proportions by arm of those who had placebo/Triazavirin withheld permanently.
To determine the proportion of patients who stop taking either placebo/Triazavirin | 1 month per patient
  We will report on tolerability by comparing the proportions by arm who had placebo/Triazavirin withheld permanently.

CONTACTS AND LOCATIONS:
Overall Officials: Neil A Martinson, MBChB, Principal Investigator — Perinatl HIV Research Unit CEO
Locations (1):
- The Perinatal HIV Research Unit - Matlosana, Klerksdorp, North West, South Africa

IPD SHARING:
Plan to Share IPD: No